CLINICAL TRIAL: NCT05987995
Title: Is it Safe to do Endometrial Injury in the Same ICSI Cycle: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0105711
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-09

CONDITIONS: Infertility
Keywords: Endometrial injury; ICSI; infertility; pregnancy rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometrial injury group (Experimental): Endometrial injury was done on day 3-5 of stimulation, just after the cessation of menstruation. After the insertion of a vaginal speculum, the cervix was cleaned using a sterile saline solution. A pipelle endometrial sampler was introduced gently into the uterine cavity. The inner piston of the catheter was withdrawn to create suction, and injury (scratching) of the endometrium was done by moving the pipelle catheter up and down within the uterine cavity. The obtained tissues were seen in a transparent tube. If no tissues were seen in the tube, the procedure was repeated.
  Interventions: Procedure: Endometrial injury
- Control group (No Intervention): no thing is done for this group

INTERVENTIONS:
Procedure: Endometrial injury — A pipelle endometrial sampler was introduced gently into the uterine cavity. The inner piston of the catheter was withdrawn to create suction, and injury (scratching) of the endometrium was done by moving the pipelle catheter up and down within the uterine cavity
  Arms: Endometrial injury group

SUMMARY:
Endometrial injury is one of the interventions suggested to improve the endometrial receptivity by enhancing the decidualization process, and so increasing the pregnancy rate

DETAILED DESCRIPTION:
In assisted reproductive techniques , specially ICSI, several approaches have been put forward to improve the endometrium, including endometrial injection of granulocyte colony-stimulating factor or platelet-rich plasma. Endometrial injury is one of the interventions suggested to improve the endometrial receptivity.

Endometrial injury, also known as endometrial scratching, is the intentional damage of the endometrium, usually using a pipelle, aiming at increasing the implantation rate. The exact mechanism of action is still vague ,many hypotheses have been advocated, including enhanced decidualization, which is stimulated by the local injury. Moreover, endometrial injury stimulates an inflammatory response, which in turn adjusts gene expression.

The value of endometrial injury is a controversial issue, there is no agreement on the exact time to perform endometrial scratching, so in the current study, we investigated the safety and efficacy of performing endometrial injury in the follicular phase of the same ICSI cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age <40 year.
* BMI 20-35 kg/m2.

Exclusion Criteria:

* Age >40 year
* BMI > 35
* Uterine cavity abnormalities
* poor quality embryos
* Poor responders
* Diagnosed sever endometriosis
* Sever male factor
* Declined to participate

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — infertile females that seeking pregnancy
Enrollment: 60 (Actual)
Dates: Start 2022-09-11 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 15 days after HCG administration
  Quantitative beta HCG test is done

CONTACTS AND LOCATIONS:
Locations (1):
- Tamer, Alexandria, Egypt